CLINICAL TRIAL: NCT03286764
Title: Use of Peppermint Oil During Screening Colonoscopy to Improve Visibility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Kevin C. Ruff, M.D., PI, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 14-006242
Record Dates: First submitted 2017-09-15; First posted 2017-09-18 (Actual); Last update posted 2020-04-03 (Actual); Status verified 2020-04

CONDITIONS: Enhancement of the ADR During Colonoscopy
MeSH Terms: interventions — peppermint oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Distilled water spray as a placebo during Colonoscopy
  Interventions: Other: Distilled water
- Peppermint Oil (Experimental): Peppermint Oil spray during Colonoscopy
  Interventions: Other: Peppermint Oil

INTERVENTIONS:
Other: Peppermint Oil
  Arms: Peppermint Oil
Other: Distilled water — Distilled water spray as a placebo during Colonoscopy
  Arms: Placebo

SUMMARY:
The investigators hypothesize that spraying peppermint oil containing L-menthol onto the colonic mucosa during colonoscopy will relax smooth muscle allowing better colonic visualization.

ELIGIBILITY:
Inclusion Criteria:

* Screening colonoscopy
* Age 50 years and older
* Able to give consent

Exclusion Criteria:

* No consent obtained or adult lacking capacity to consent
* Do not reach cecum on colonoscopy
* Renal impairment (defined as CrCl <30 ml/min)
* Allergy to study peppermint oil solution
* History of colon resection
* Inflammatory bowel disease
* Known colorectal neoplasia
* Non-correctable coagulopathy
* Pregnancy or lactating
* Prisoners

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2016-11; Primary Completion 2019-09-10 (Actual); Study Completion 2019-09-10 (Actual)

PRIMARY OUTCOMES:
Determination of Adenoma Detection Rate during Colonoscopy Procedure | 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Kevin C Ruff, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials